CLINICAL TRIAL: NCT02914015
Title: Ultrasound-guided Continous Quadratus Lumborum Block: Effect on Acute Pain and Quality of Recovery After Hepatic Surgery With Right Subcostal Incision
Brief Title: Continous Quadratus Lumborum Block for Hepatic Surgery With Right Subcostal Incision
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: we change the study protocol
Sponsor: Cui Xulei (Other)
Responsible Party: Sponsor-Investigator, Cui Xulei, Attending Physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CXL4
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Hepatectomy; Analgesia; Nerve Block
MeSH Terms: conditions — Agnosia | interventions — Catheterization; Ropivacaine; isopropyl cyanoacrylate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous QLB+postoperative IPCA (Experimental): Single-injection of QLB (quadratus lumborum block) is given preoperatively followed with continuous infusion+ postoperative IPCA (intravenous patient control analgesia)
  Interventions: Procedure: Continous QLB (quadratus lumborum block); Device: Philip CX50 Ultrasound Scanner; Drug: Ropivacaine; Drug: Morphine given as IPCA
- IPCA (Active Comparator): Postoperative IPCA (intravenous patient control analgesia) is given alone
  Interventions: Drug: Morphine given as IPCA

INTERVENTIONS:
Procedure: Continous QLB (quadratus lumborum block) — Inject local anesthetics in between quadratus lumborum and psoas major muscle with catheter insertion and continuous local infusion
  Other Names: Inject local anesthetics in between quadratus lumborum and psoas major muscle with catheter insertion and continuous local infusion
  Arms: Continuous QLB+postoperative IPCA
Device: Philip CX50 Ultrasound Scanner — The curved (C1-5) probe of Philip CX 50 Ultrasound Scanner is used for scan
  Arms: Continuous QLB+postoperative IPCA
Drug: Ropivacaine — * 0.6ml/kg 0.5% ropivacaine with 1:200,000 adrenaline given immediately after the correct position of the tip of the needle has been verified.
  * followed with 0.2% ropivacaine infusion at a rate of 0.125ml/kg/h given through the catheter inserted in between the quadratus lumborum muscle and psoas major muscle.
  Arms: Continuous QLB+postoperative IPCA
Drug: Morphine given as IPCA — Bolus: 1-2mg, lock time: 10min, 1h limitation: 5-10mg. without background infusion.

SUMMARY:
This prospective, randomized study, control study aims to compare the analgesic effect, opioids consumption, quality of recovery, length of hospital stay and et al. between unilateral continuous quadratus lumborum block (QLB) and intravenous patient-controlled analgesia (IPCA) alone in patients undergoing hepatectomy with right J-shape subcostal incision.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo hepatectomy with right J-shape subcostal incision
* Informed consent

Exclusion Criteria:

* A known allergy to the drugs being used
* Coagulopathy, on anticoagulants
* Analgesics intake, history of substance abuse
* Participating in the investigation of another experimental agent
* Inability to properly describe postoperative pain to investigators (eg, language barrier, neuropsychiatric disorder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Cumulative morphine consumption | at 24 postoperative hours

SECONDARY OUTCOMES:
The pain scores determined by the numeric rating scale (NRS, 0-10) | At 0, 2,4, 8, 12, 24 ,48,72 hours and 7 day after the surgery
Nausea and Vomiting score | At 0, 2,4, 8, 12, 24 and 48 hours after the surgery
Pruritus score | At 0, 2,4, 8, 12, 24 and 48 hours after the surgery
Ambulation time | within the 7 days after surgery
Time of recovery of bowl movement | within the 7 days after surgery
Quality of recovery | 3 days and 7 days after surgery
  use the self-assessment 11 item QoR scale to assess the patient's recovery quality
Patient satisfaction with anesthesia | 48 hours after surgery
  use the Chinese version Bauer questionnaire to assess the patient satisfaction with anesthesia
Postoperative hospital length of stay | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, MD., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Xulei CUI, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No